CLINICAL TRIAL: NCT03732612
Title: The Role of Inflammation in Vascular Disease (Inflammationens Roll i kärlsjukdom)
Brief Title: Inflammation in Vascular Disease
Acronym: REBEL
Status: Recruiting | Type: Observational
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Other Study IDs: 660-18
Record Dates: First submitted 2018-11-05; First posted 2018-11-06 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-05

CONDITIONS: Vascular Diseases; Atherosclerosis
MeSH Terms: conditions — Vascular Diseases; Atherosclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Vascular tissue.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control patients: Control patients (n=20): In individuals undergoing vascular surgery that is not associated with vascular disease (e.g. knee replacement surgery, trauma, etc), a piece of healthy vessel must sometimes be removed in order to facilitate the surgical process. The vessel biopsies from this group will be categorized as "healthy vessels" in our study.
- Study patients: Study patients (n=150): In individuals undergoing vascular surgery associated with peripheral arterial diseases, aneurysm and/or other manifestations of atherosclerosis, vascular tissue is sometimes excised to facilitate the surgery. Biopsies from these individuals will be categorized as "vessels with vascular dysfunction".

SUMMARY:
Increasing evidence suggests that systemic low-grade inflammation may be a driving force of cardiometabolic complications, such as vascular dysfunction, atherosclerosis and ischemic heart disease. Thus, we will investigate the role of inflammation in cardiovascular disease.

DETAILED DESCRIPTION:
Vascular reconstruction surgeries usually require a small piece of the vessel wall to be excised. The excised vessel is generally discarded as medical waste: however, for patients participating in the study, the excised tissue will be placed in saline and collected for research use.

Tissue collected from individuals undergoing vascular surgery associated with peripheral arterial diseases, aneurysm and/or other manifestations of atherosclerosis, vascular tissue will be cultured ex vivo in the presence or absence of therapeutic agents, to determine if these attenuate the inflammation associated with the atherosclerotic phenotype. Furthermore, the protocol will also be carried out using vascular tissue from control patients, which have undergone vascular surgery that is not associated with vascular disease (e.g. knee replacement surgery, trauma, etc).

ELIGIBILITY:
Inclusion Criteria:

* Patient is planned to undergo vascular surgery.
* Signed informed consent has been obtained from the patient.

Exclusion Criteria:

* Patient has difficulty to understand information.
* Patients under 18 years of age.
* Patients participating in any drug-related study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Consecutive patients planned for vascular reconstruction surgery at our center.
Sampling Method: Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2019-09-02 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Inflammatory status | 2019-2024
  The inflammatory status will be studied in patients with atherosclerotic disease.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Boren, MD, PhD, Study Director — The University of Gothenburg
Locations (1):
- University of Gothenburg, Gothenburg, Vastragotaland, Sweden